CLINICAL TRIAL: NCT01716416
Title: A Phase I Trial of Pazopanib Suspension Plus Cetuximab in Patients With Incurable Head and Neck Squamous Cell Carcinoma
Brief Title: Pazopanib Plus Cetuximab for Incurable Head and Neck Squamous Cell Carcinoma (HNSCC)
Acronym: HNSCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201211110
Record Dates: First submitted 2012-10-24; First posted 2012-10-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pazopanib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level 1 (Experimental): Pazopanib 200 mg PO QD
  Cetuximab 400 mg/m^2 (cycle 1 week 1 only) followed by weekly maintenance doses of 250 mg/m^2
  Interventions: Drug: Pazopanib; Drug: Cetuximab
- Dose Level 2 (Experimental): Pazopanib 400 mg PO QD
  Cetuximab 400 mg/m^2 (cycle 1 week 1 only) followed by weekly maintenance doses of 250 mg/m^2
  Interventions: Drug: Pazopanib; Drug: Cetuximab
- Dose Level 3 (Experimental): Pazopanib 600 mg PO QD
  Cetuximab 400 mg/m^2 (cycle 1 week 1 only) followed by weekly maintenance doses of 250 mg/m^2
  Interventions: Drug: Pazopanib; Drug: Cetuximab
- Dose Level 4 (Experimental): Pazopanib 800 mg PO QD
  Cetuximab 400 mg/m^2 (cycle 1 week 1 only) followed by weekly maintenance doses of 250 mg/m^2
  Interventions: Drug: Pazopanib; Drug: Cetuximab
- Part 2 Dose (Experimental): Pazopanib (dose to be determined in Part 1 of study) mg PO QD
  Cetuximab 400 mg/m^2 (cycle 1 week 1 only) followed by weekly maintenance doses of 250 mg/m^2
  Interventions: Drug: Pazopanib; Drug: Cetuximab

INTERVENTIONS:
Drug: Pazopanib
  Other Names: Votrient®
Drug: Cetuximab
  Other Names: Erbitux®

SUMMARY:
This phase I trial studies the side effects and best dose of pazopanib hydrochloride (pazopanib) when given together with cetuximab in treating patients with incurable recurrent or metastatic head and neck cancer. Pazopanib may stop the growth of cancer by blocking blood flow to the tumor. Pazopanib may also block some of the enzymes needed for cell growth. Cetuximab is a monoclonal antibody that blocks the ability of some tumor cells to grow and spread. Giving pazopanib with cetuximab may provide a more effective treatment for patients with advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed diagnosis of incurable metastatic or recurrent head and neck squamous cell carcinoma
* Patient must have measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm with CT scan, as ≥20 mm by chest x-ray, or ≥10 mm with calipers by clinical exam (Expanded Cohort only; patients without measurable disease by RECIST 1.1 criteria but with evaluable disease will be eligible for the dose-finding phase).
* Patient must be ≥ 18 years of age.
* Patient must have an ECOG performance status 0-1
* Patient must have normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * INR ≤ 1.2 x IULN; patients receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation
  * aPTT ≤ 1.2 x IULN
  * Corrected QT interval (QTc) < 480 msecs
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT) ≤ 2.5 x IULN and ALT(SGPT) ≤ 2.5 x IULN
  * Creatinine ≤ 1.5 mg/dL OR Creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with creatinine levels > 1.5 mg/dL
  * Urine protein to creatinine ratio (UPC) < 1; if UPC ≥ 1, then a 24-hour urine protein must be assessed; patients must have a 24-hour urine protein value < 1 g to be eligible
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) beginning 14 days prior to first dose of pazopanib, through the dosing period, and for at least 28 days after the last dose of pazopanib.
* Patient must be able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* For the expanded cohort only, patient must not have had prior therapy with an EGFR-specific monoclonal antibody or EGFR-specific TKI for treatment of incurable HNSCC. Prior therapy with an EGFR-specific monoclonal antibody as part of the definitive treatment of curable HNSCC is acceptable if this occurred more than 3 months prior to study enrollment. For the dose-finding cohorts, prior EGFR-specific therapy in the incurable setting is allowed.
* Patient must not have had radiation therapy, minor surgery, or tumor embolization with 14 days prior to the first dose of pazopanib.
* Patient must not have had chemotherapy, immunotherapy, biologic therapy, hormonal therapy, or investigational therapy within 14 days or 5 half-lives of the drug prior to the first dose of pazopanib. For patients enrolling in the phase I portion of this study, this requirement does not apply to prior treatment with cetuximab.
* Patient must not have prior major surgery, trauma, presence of any non-healing wound, fracture, or ulcer within 28 days prior to first dose of study drug.
* Patient must not have a history of other malignancy ≤ 2 years previous with the exception of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma.
* Patient must not be receiving any medication that is a strong CYP3A4 inhibitor beginning 14 days prior to first dose of study drug. Strong CYP3A4 inhibitors include (but are not limited to): antibiotics such as clarithromycin, telithromycin, troleandromycin; protease inhibitors such as ritonavir, indinavir, saquinavir, nelfinavir, lopinavir; antifungals such as itraconazole, ketoconazole, voriconazole; and antidepressants such as nefazodone.
* Patient must not be receiving any other investigational agents.
* Patient must not be experiencing any ongoing toxicity from prior anti-cancer therapy that is > grade 1 or that is progressing in severity, except alopecia.
* Patient must not have a history of or clinical evidence of central nervous system metastases or leptomeningeal carcinomatosis, except for individuals who have had previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medications for 6 months prior to first dose of pazopanib.
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib, cetuximab, or other agents used in the study.
* Patient must not have any clinically significant gastrointestinal abnormality that may increase the risk of GI bleeding including, but not limited to, active peptic ulcer disease, known intraluminal metastatic lesions with risk of bleeding, inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease), other GI conditions with increased risk of perforation, history of abdominal fistula or GI perforation or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Patient must not have any clinically significant abnormality that may affect absorption of investigational product including, but not limited to, malabsorption syndrome or major resection of the stomach or small bowel.
* Patient must not have an uncontrolled intercurrent illness within the 6 months prior to study entry including, but not limited to, ongoing or active infection, Class III or IV congestive heart failure (as defined by the New York Heart Association (NYHA)), unstable angina pectoris, cardiac arrhythmia, myocardial infarction, cardiac angioplasty or stenting, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not have poorly controlled hypertension (defined as systolic blood pressure of ≥ 140 mmHg or diastolic blood pressure of ≥ 90 mmHg). Initiation or adjustment of antihypertensive medications is permitted prior to study entry. Blood pressure must be re-assessed on two occasions that are separated by a minimum of one hour; on each of these occasions, the mean (of 3 readings) from each assessment must be < 140/90 mmHg for a patient to be eligible for this study.
* Patient must not have a history of cerebrovascular accident including transient ischemic attack within the past 6 months. Patients with recent deep venous thrombosis or pulmonary embolism who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible as long as INR is stable.
* Patient must not have evidence of active bleeding or bleeding diathesis.
* Patient must not have any known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
* Patient must not experience hemoptysis in excess of 2.5 mL within 8 weeks prior to the first dose of pazopanib.
* Patient must not be pregnant and/or breastfeeding. Patient must have a negative serum pregnancy test within 14 days of study entry.
* Patient must not be known to be HIV-positive on combination antiretroviral because of the potential for pharmacokinetic interactions with pazopanib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose (MTD) of pazopanib suspension when combined with fixed dose cetuximab in patients with incurable HNSCC. | 9 weeks (completion of all patients in part 1 of study through 1st cycle)

SECONDARY OUTCOMES:
Early Adverse events | 8 weeks
  Graded by NCI-CTC criteria version 4 and described in a frequency distribution analysis for the first 8 weeks of pazopanib and cetuximab
Late adverse events | Weeks 8 through 16
  Graded by NCI-CTC criteria version 4 and described in a frequency distribution analysis for subsequent interval (after first 8 weeks of therapy) of receiving pazopanib and cetuximab
Anatomic tumor response | 8 weeks
  Assessed by CT and clinical exam
Overall metabolic response | 8 weeks
  Assessed by FDG-PET
Overall response rate | 8 weeks
  CR+PR
Duration of overall response | 8 weeks
  Time from CR or PR until relapse
Best overall response rates in patients treated with MTD | 8 weeks
  According to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adkins D, Mehan P, Ley J, Siegel MJ, Siegel BA, Dehdashti F, Jiang X, Salama NN, Trinkaus K, Oppelt P. Pazopanib plus cetuximab in recurrent or metastatic head and neck squamous cell carcinoma: an open-label, phase 1b and expansion study. Lancet Oncol. 2018 Aug;19(8):1082-1093. doi: 10.1016/S1470-2045(18)30350-4. Epub 2018 Jul 11. PMID 30001987
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu